CLINICAL TRIAL: NCT04849884
Title: A Prospective, Multi-Center, Post-Market Clinical Study to Evaluate the Performance of the CORI™ KNEE TENSIONER as an Accessory to the CORI™ Surgical System in Total Knee Arthroplasty Procedures.
Brief Title: To Evaluate the Performance of the CORI™ KNEE TENSIONER as an Accessory to the CORI™ Surgical System.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CORI TENSIONER.2020.04
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Arthroplasty; Replacement; Knee
Keywords: Total Knee Arthroplasty (TKA); Robotic; CORI™ KNEE TENSIONER; CORI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- CORI TENSIONER (Experimental): Subjects having a robotic TKA procedure with the CORI Surgical System, including the use of the CORI™ KNEE TENSIONER accessory.
  Interventions: Device: CORI™ KNEE TENSIONER

INTERVENTIONS:
Device: CORI™ KNEE TENSIONER — Robotic TKA procedure with the REAL INTELLIGENCE™ CORI™ Surgical System including the use of the CORI™ KNEE TENSIONER accessory.

SUMMARY:
To evaluate the performance of the CORI™ KNEE TENSIONER as an accessory to the CORI™ Surgical System.

DETAILED DESCRIPTION:
This is a post-market, prospective, multicenter, open-label study evaluating the performance of the CORI™ KNEE TENSIONER as an accessory to the CORI™ Surgical System at approximately 4 centers across the United States. Ninety (90) patients eligible for a robotic-assisted TKA procedure with the CORI™ Surgical System will be followed for approximately 12 months.

The CORI™ KNEE TENSIONER is an accessory to REAL INTELLIGENCE™ CORI™ Surgical System. The TENSIONER may assist the surgeon in providing consistent varus and valgus stress during gap assessment before making any bony resections. The TENSIONER communicates directly with CORI software, providing automated data collection.

The primary objective is to evaluate the performance of the CORI™ KNEE TENSIONER as an accessory to the CORI™ Surgical System by assessing patient satisfaction with the EQ-5D-5L VAS.

ELIGIBILITY:
Inclusion Criteria:

1. Subject agrees to consent to the study by signing the Independent Review Board (IRB) approved ICF.
2. Subject is eighteen (18) years old or older.
3. Subject is willing and able to attend all study follow-up visits for up to one (1) year postoperatively (as defined in the study protocol and ICF).
4. Subject can read, understand, and communicate responses to Patient Reported Outcome Measures (PROMs).
5. Subject is suitable for the CORI™ Surgical System.
6. Subject requires a cemented TKA as a primary indication due to any of the following conditions:

   * Degenerative joint disease, including osteoarthritis
   * Rheumatoid arthritis.
   * Avascular necrosis.
   * Requires correction of functional deformity
   * Requires treatment of fractures that were unmanageable using other techniques.

Exclusion Criteria:

1. Contraindications or hypersensitivity to the use of the CORI™ Surgical System per the IFU.
2. Participation in the treatment period of another clinical trial within thirty (30) days of the Pre-Operative Visit, or during the study.
3. Women who are pregnant, nursing, or of child-bearing potential who are not utilizing birth control measures.
4. Subjects who are non-English speaking.
5. Any subject that meets the definition of a Vulnerable Subject per ISO 14155.
6. Subjects who have participated previously in this clinical trial
7. Subjects with a history of poor compliance with medical treatment.
8. Subject needs a CORI™ Surgical System TKA on the index joint as a revision for a previously failed surgery, or need for complex implants, or any other implant than a standard TKA (e.g., stems, augments, or custom-made devices).
9. Subject has been diagnosed with post-traumatic arthritis
10. Subject needs a bilateral TKA.
11. Subject has active infection or sepsis (treated or untreated)
12. Subject is morbidly obese with a body mass index (BMI) greater than 40.
13. Subjects with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study. This includes:

    * Advanced osteoarthritis
    * Joint disease
    * Paget's or Charcot's disease
    * Vascular insufficiency
    * Muscular atrophy
    * Uncontrolled diabetes
    * Moderate to severe renal insufficiency
    * Neuromuscular disease
    * Mental illness or mental retardation
    * Drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-10 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Life: EuroQol 5-Dimension 5-Level Visual Analogue Scale (EQ-5D-5L VAS) at 12 months | 12 months
  The VAS records the subject's self-rated health on a vertical visual analogue scale. The endpoints on the scale are labelled "The best health you can imagine" and "The worst health you can imagine". Participants indicate a numerical value from 1-100 where 0 is the worst imaginable health state and 100 is the best imaginable health state. The VAS can be used as a quantitative measure of health outcome as judged by the individual respondents.

SECONDARY OUTCOMES:
Quality of Life: EuroQol 5-Dimension 5-Level Visual Analogue Scale (EQ-5D-5L VAS) pre-operative, 6 weeks, and 6 months | pre-operative, 6 weeks, and 6 months
  The VAS records the subject's self-rated health on a vertical visual analogue scale. The endpoints on the scale are labelled "The best health you can imagine" and "The worst health you can imagine". Participants indicate a numerical value from 1-100 where 0 is the worst imaginable health state and 100 is the best imaginable health state. The VAS can be used as a quantitative measure of health outcome as judged by the individual respondents.
Quality of Life (EQ-5D-5L Index score) | Pre-operative, 6 weeks, 6 months, and 12 months
  The EQ-5D-5L will be collected at the preoperative visit and at the 6-week, 6-month,& 12-month Follow-Up Visits.
  The descriptive system is used to describe the subject's health state & consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels to choose the most appropriate answer: no problems, slight problems, moderate problems, severe problems, and extreme problems. The subject is asked to indicate his/her health state by marking the most appropriate statement in each of the five areas. Responses are coded as single-digit numbers expressing the severity level selected in each dimension. For instance, 'slight problems' (e.g. 'I have slight problems in walking about') is always coded as '2'. The digits for the 5 dimensions are combined in a 5-digit code. The EQ- 5D-5L index value is derived by using the vendor supplied calculator to convert each 5-digit EQ-5D-5L profile. A higher number is a better outcome.
2011 Knee Society Score (KSS) | Pre-operative, 6 weeks, 6 months, and 12 months
  The 2011 KSS will be collected at the preoperative visit and at the 6-week, 6-month, and 12-month Follow-Up Visits.
  The KSS is a validated tool that combines an objective physician-derived component with a subjective subject-derived component and consists of 4 separate sub-scales:
  1. An "Objective" Knee Score (seven items: 100 points)
  2. A Patient Satisfaction Score (five items: 40 points)
  3. A Patient Expectation Score (three items: 15 points)
  4. A Functional Knee Score (19 items: 100 points)
  The Functional Knee Score is derived from assessments of walking and standing, standard activities, advanced activities, and discretionary activities. A higher number is a better outcome.

OTHER OUTCOMES:
Medial-to-lateral balance measurements at 0/10°, 30°, 60°, and 90° flexion. | During surgical procedure
  Gap planning measurements will be defined as the medial-to-lateral balance measurements at 0/10°, 30°, 60°, and 90° flexion.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Hospital for Special Surgery, New York, New York
  - OrthoNeuro, New Albany, Ohio
  - University of Pittsburgh, Magee, Pittsburgh, Pennsylvania
  - Memorial Medical Center, Ashland, Wisconsin

IPD SHARING:
Plan to Share IPD: No